CLINICAL TRIAL: NCT04707599
Title: Reducing the Rate of Missed Appointments in an Outpatient Substance Use Treatment Clinic in Norway
Brief Title: Telephone Reminder to Increase Appointment Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 005004 - 2014/2225
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2021-01

CONDITIONS: Reminder Systems; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental with an OFF-ON design
Who Masked: Participant
Masking Description: The aim of the study was presented to all participants (to examine dropout/ retention from treatment), but patients were blinded to information about the phase comparison (i.e., that there was a pretreatment telephone Call from therapist in one phase and not in the other).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFF intervention (No Intervention): No reminder plus (telephone reminder from therapist) but standard test message reminder (SMS) from second admission
- ON intervention (Experimental): Reminder plus (telephone reminder from therapist) AND standard test message reminder (SMS) from second admission
  Interventions: Other: Reminder plus (telephone call from therapist)

INTERVENTIONS:
Other: Reminder plus (telephone call from therapist) — Reminder plus (telephone call from therapist)
  Arms: ON intervention

SUMMARY:
Missed appointments to outpatient substance use treatment are common and costly and can have a negative effect on the health of patients.

In this quasi-experimental study, the investigators used an on-off design to examine whether a reminder "plus" intervention (telephone call from therapist before first appointment) would increase attendance and improve cancellation and rebooking practices. Secondary outcomes included satisfaction with treatment and intention to complete the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patient
* > 18 years
* Diagnosis: Substance related disorder

Exclusion Criteria:

* Patients who are unable to understand or score the survey due to cognitive or language barriers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Attendance rate | Up to 10 treatment sessions, estimated average timeframe = 3 months
  Attendance rate at first admission and during 10 outpatient sessions

SECONDARY OUTCOMES:
Dropout rate | Up to 10 treatment sessions, estimated average timeframe = 3 months
  Dropout rate within 10 sessions - measured as formal discharge and/or "technical discharge" (3x no-shows)
Cancellation / rebooking rate | Up to 10 treatment sessions, estimated average timeframe = 3 months
  Examine difference in cancellation / rebooking rate between the two conditions. Data was collected from administrative patient records.

OTHER OUTCOMES:
Treatment satisfaction | First week
  Treatment satisfaction - measured with the Session Rating Scale (scale 0 - 40, higher scores means higher satisfaction)
Intention to complete treatment | First week
  Intention to complete treatment program. Self-developed measured based on the Theory of Planned Behavior. Scale 1 - 7, higher scores means higher intention to Complete treatment).

CONTACTS AND LOCATIONS:
Overall Officials: John-Kåre Vederhus, PhD, Principal Investigator — Sørlandet Hospital
Locations (2):
- Norway (2):
  - Addiction Unit - Sørlandet Hospital, Arendal, Agder
  - Addiction Unit - Sørlandet Hospital, Kristiansand, Agder

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallefoss LJ, Gabrielsen KB, Haugland SH, Clausen T, Vederhus JK. Effects of a brief pre-admission telephone reminder on no-show and dropout rates in substance use disorder treatment: a quasi-experimental study. Subst Abuse Treat Prev Policy. 2022 Aug 23;17(1):61. doi: 10.1186/s13011-022-00489-9. PMID 35999633